CLINICAL TRIAL: NCT05019534
Title: A Phase I Study on Tolerance and Safety of Vemurafenib Film-coated Tablets, Cetuximab Solution for Infusion and Camrelizumab Protocol(VCC) in the After Line Therapy of BRAF V600E Mutation/MSS Metastatic Colorectal Cancer
Brief Title: Tolerability and Safety of Vemurafenib, Cetuximab Combined With Camrelizumab for BRAF V600E-mutated /MSS Metastatic Colorectal Cancer
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: West China Hospital (Other)
Responsible Party: Principal Investigator, Meng Qiu, Clinical Professor, West China Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ChiECRCT20210210
Record Dates: First submitted 2021-08-05; First posted 2021-08-25 (Actual); Last update posted 2022-05-19 (Actual); Status verified 2022-05

CONDITIONS: BRAF V600E-mutated /MSS Metastatic Colorectal Cancer; Vemurafenib (BRAFi) Plus Cetuximab (EGFRi) Combined With PD-1 Monoclonal Antibody
MeSH Terms: interventions — Vemurafenib; Cetuximab; camrelizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Vemurafenib, Cetuximab Combined With Camrelizumab (VCC) (Experimental): Cetuximab and Camrelizumab in the fixed dose Vemurafenib have two dose groups: 960mg qd or 960mg bid
  Interventions: Drug: Vemurafenib Oral Tablet [Zelboraf]; Drug: Cetuximab Injection [Erbitux]; Drug: Camrelizumab

INTERVENTIONS:
Drug: Vemurafenib Oral Tablet [Zelboraf] — Vemurafenib 960mg qd or 960mg bid (2 cohorts)
  Other Names: Zelboraf
Drug: Cetuximab Injection [Erbitux] — Cetuximab 500mg/m2 Q2W
  Other Names: Erbitux
Drug: Camrelizumab — Camrelizumab 200mg Q2W

SUMMARY:
BRAF mutation exists in about 10-12% of colorectal cancer, among which BRAF V600E mutation is the most common type, which is an important biomarker for predicting the prognosis and precise treatment efficacy of metastatic colorectal cancer (mCRC). The prognosis of metastatic colorectal cancer with BRAF V600E mutation is very poor, with OS of about 6-9 months. Previous studies have shown that single anti-BRAF inhibitor are ineffective, while multi-target inhibitions of Ras-Raf -MEK pathway is a possible effective strategy for BRAF V600E-mutant mCRC. Currently, the proven effective regimens include the VIC regimen (Vemurafenib + cetuximab + Irinotecan) and BEACON regimen (Encorafenib+ cetuximab +/- Binimetinib) from the SWOGS1406 study. Furthermore, BRAF inhibitor +MEK inhibitor combined with PD-1 monoclonal antibody has been shown to be an effective strategy in BRAF V600E-mutant malignant melanoma, which promote the study of the regimens for the treatment of BRAF V600E-mutant mCRC. Increasing basic and clinical studies have shown that cetuximab has ADCC effect, induces immunogenic cell death, promotes immune cell infiltration and other immunomodulatory effects, and has a synergistic effect with PD-1 monoclonal antibody in colorectal cancer. Based on those theories, we conducted the phase I study to explore the safety and preliminary efficacy of the regimen of Vemurafenib (BRAFi) plus cetuximab (EGFRi) combined with PD-1 monoclonal antibody in BRAF V600E-mutant /MSS type mCRC.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female ≥ 18 years of age
2. Eastern Cooperative Oncology Group (ECOG) Performance Status of 0-2
3. Participants must have histologically or cytologically confirmed diagnosis of adenocarcinoma of the colon or rectum, with clinical confirmation of unresectable and/or metastatic disease that is measurable according to Response Evaluation Criteria in Solid Tumors (RECIST 1.1) criteria
4. Presence of BRAF V600E in tumor tissue determined by local assay at any time prior to screening and confirmed by central laboratory. And confirmation of MSS or pMMR status from immunohistochemistry or PCR or NGS;
5. Prior treatment with at least one systemic treatment (chemotherapy or target therapy) for mCRC, and prior treatment did not include cetuximab
6. Adequate organ and marrow function:

   * ①Hemoglobin (Hb) ≥ 90 g/L；Platelets (PLT) ≥ 75 x 10^9/L；Neutrophil ≥1.5 x 10^9/L
   * ②Total bilirubin ≤ 1.5 x upper limit of normal (ULN)；Aspartate aminotransferase (AST) ≤3 x ULN ；Alanine aminotransferase (ALT) ≤3 x ULN
   * ③Serum creatinine ≤ 1.5 x ULN, or calculated creatinine clearance (determined as per Cockcroft-Gault) ≥ 50 mL/min at screening
   * ④INR, APTT, and PT≤ 1.5 x ULN
   * ⑤Serum albumin≥ 28 g/L
   * ⑥ECG showed no evident abnormality
7. Written informed consent

Exclusion Criteria:

1. Known hypersensitivity or contraindication to any component of cetuximab or PD-1 monoclonal antibody or macromolecular protein reagent.
2. A history of other malignancies with a disease-free survival of less than 5 years, with the following exceptions: adequately treated basal or squamous cell skin cancer, carcinoma in-situ of the cervix, and gastrointestinal tumors treated curatively with endoscopic mucosectomy;
3. Any active autoimmune disease or a history of autoimmune disease
4. Use of immunosuppressive medications or glucocorticoid therapy ≤2 weeks prior to entry
5. Uncontrolled active infection requiring antibiotics
6. Known history of HIV infection or active hepatitis
7. Severe complications, including any of the following:

   * ①Massive gastrointestinal bleeding, perforation, or gastrointestinal obstruction
   * ②Symptomatic heart disease
   * ③Uncontrolled diabetes and hypertension
   * ④Uncontrolled diarrhea
8. Women who are pregnant or lactating and people who do not agree to avoid pregnancy
9. Patients with serious psychiatric that may interfere treatment.
10. Other conditions which are inappropriate to participate in the study confirmed by investigators.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Estimated)
Dates: Start 2021-08-15 (Actual); Primary Completion 2022-08-01 (Estimated); Study Completion 2022-12-01 (Estimated)

PRIMARY OUTCOMES:
Evaluate tolerability and safety and identify the recommended Phase 2 dose(RP2D) | Subjects will be treated and observed for dose-limiting toxicity(DLT) through the end of the first cycle (Days 1-28)

SECONDARY OUTCOMES:
Object Response Rate (ORR) | up to 24 weeks
  Rate of patients with partial or complete response according to modified RECIST criteria.
Disease Control Rate (DCR) | up to 24 weeks
  the proportion of patients who had a best response rating of complete response, partial response, or stable disease according to modified RECIST
Progression Free Survival (PFS) | up to 1 year
  Progression free survival (Medium, Kaplan-Meier-estimation, ITT- population)
Overall Survival (OS) | up to 3 year
  Overall survival (Kaplan-Meier-estimation, ITT- population)
Preliminary efficacy | up to 1 year
  Evaluation of preliminary efficacyaccording to RECIST 1.1

CONTACTS AND LOCATIONS:
Locations (1):
- Sichuan University West China Hospital, Chengdu, Sichuan, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Wei GX, Zhou YW, Cao P, Leng WB, Wang L, Tang J, Qiu M. Vemurafenib, cetuximab and camrelizumab in BRAF V600E-mutated/MSS metastatic colorectal cancer. J Transl Med. 2025 Nov 12;23(1):1274. doi: 10.1186/s12967-025-07312-6. PMID 41225509